

## Empirical testing of a widely available insurance-based monetary incentive program for exercise: A randomized trial

**NCT Number: N/A** 

ID: R01 CA262894

January 4, 2023



## BROWN UNIVERSITY CONSENT FOR RESEARCH PARTICIPATION

## **Exercise for Good**

[Version 2, 12/12/2022]

You are invited to take part in a Brown University research study. Your participation is voluntary.

- RESEARCHERS: You are being asked to take part in a research study conducted by Drs. David Williams and Omar Galárraga. Dr. Williams has a Ph.D. in Psychology and is a Professor of Behavioral and Social Sciences at the Brown University School of Public Health. Dr. Galárraga has a Ph.D. in Health Economics and is an Associate Professor of Health Services, Policy, and Practice at the Brown University School of Public Health. To contact the study staff call 401-XXX-XXXX or email exercise4good@brown.edu.
- PURPOSE: This study is about seeing if a monetary incentive will help you develop a more physically active lifestyle by attending the YMCA more frequently. You are being asked to be in this study because you are a current member of the Greater Providence YMCAs.
- PROCEDURES: You will be asked to complete questionnaires and wear an Actigraph activity monitor at the beginning of the study and at 3-month intervals (5 times total) during the 12-month study. We will also be monitoring your facility usage (e.g. the number of times you use any of the Greater Providence YMCA branches) at the YMCA. This information is used for research purposes only to evaluate the study. We cannot see what you did at the YMCA, or how long you were there, only the date and time you checked into the YMCA, and the branch you checked into. When you signed up for a YMCA membership, one of the terms in the YMCA membership agreement is that they electronically track your facility usage when you swipe your membership card to attend the YMCA. Lastly, if you are randomly assigned to one of the incentive conditions, you will be asked to mail us a copy of your YMCA attendance records and payment receipts to receive the incentive.
- TIME INVOLVED: The study will take 5-7 hours of your time over a period of 12 months, as well as the amount of time you choose to spend exercising.
- COMPENSATION: You will receive up to \$140 compensation in the form of Amazon.com gift cards for your time completing questionnaires and wearing the activity monitor. Depending on which group you are randomly assigned to, you may also earn up to an additional \$400 in the form of Visa/MasterCard gift cards as part of the incentive program.
- RISKS: You could potentially experience minor injuries or muscle sprains due to participating in an exercise program, however the likelihood of this risk is low. Previous injury or a current problem is a risk factor for future injuries. If you have or had an injury to your lower extremities



including back, hips, knees or feet, please let the study staff know. If you do become injured during the study, you should call your doctor immediately and alert the study staff. You can stop participating at any time. If you experience an illness or injury that prevents you from engaging in regular physical activity, you may be placed on a temporary medical hold until your physician clears you to continue with the study. If after you are enrolled in the study it becomes clear that you do not meet the eligibility criteria, we may ask you to withdraw from the study.

Many kinds of research involve some risk of injury. Even though the investigators are careful to prevent any harm, you might develop medical problems from being in this study. If you do have problems, the researchers will give you information that may be of help to you in getting proper medical care, if you ask for it. Brown University does not pay for medical or other costs. Signing this form does not mean that you give up any liability rights for personal injury.

- BENEFITS: You may not directly benefit from being in this research study. If you begin and continue a program of regular physical activity you may experience some health benefits.
   Regular physical activity reduces the risk of heart disease and stroke, helps control cholesterol levels, diabetes, obesity, and reduces high blood pressure for some people. Even modest levels of physical activity provide some benefit. Physical activity helps in developing endurance, joint flexibility, and muscle strength--things that are especially important as people age.
- CONFIDENTIALITY: All of your records from this study will be treated as confidential and will be protected to the fullest extent of the law. Data will be deidentified and coded with an arbitrary ID number. Participant names will only be linked to ID numbers in a password-protected file on a secure Brown University server. Data with identifying information (i.e. consent forms, contact information) will be kept separate from coded deidentified data. Any collected data will be saved on a secure Brown University server, accessible only by Dr. Williams, Galárraga and authorized research staff. Any paper data will be stored in a locked file cabinet at Brown University.

Your privacy will be maintained over Zoom video conferencing. All meetings will be secured with waiting rooms and research staff will have control over meeting settings and restrictions to ensure your privacy. We will record the audio of Zoom sessions. We will only save the audio files from the recording, we will not keep any recordings of your video. We will maintain the audio files with a participant ID number rather than your name. All audio files will be saved to a secured computer server hosted by Brown University.

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you.



The Certificate cannot be used to resist a demand for information from personnel of the United States federal or state government agency sponsoring the project and that will be used for auditing or program evaluation of agency funded projects. You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, medical care provider, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

The Certificate of Confidentiality will not be used to prevent disclosure to state or local authorities if there are any reports of child abuse, neglect, or harm to self or others.

A description of this clinical trial will be available on http://www.Clinical Trials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Finally, Brown University staff sometimes review studies like this one to make sure they are being done safely and correctly. If a review of this study takes place, your records may be examined. The reviewers will protect your confidentiality.

VOLUNTARY: You do not have to be in this study if you do not want to be. Even if you decide to be in this study, you can change your mind and stop at any time.

CONTACT INFORMATION: If you have any questions about your participation in this study, you can call Viveka at (phone #) or email exercise4good@brown.edu.

YOUR RIGHTS: If you have questions about your rights as a research participant, you can contact Brown University's Human Research Protection Program at 401-863-3050 or email them at IRB@Brown.edu.

CONSENT TO PARTICIPATE: [Online consent] Clicking the link below confirms that you have read and understood the information in this document, are over 18, and that you agree to volunteer as a research participant for this study.

You can print a copy of this form.

<include URL>